CLINICAL TRIAL: NCT05985057
Title: A Novel Approach to Antimicrobial Resistance: Machine Learning Predictions for Carbapenem-Resistant Klebsiella in ICUs
Acronym: ICU
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Volkan Alparslan, Medical Doctor, Kocaeli University
Other Study IDs: GOKAEK-2023/12.32
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Carbapenem Resistant Enterobacteriaceae Infection; Artificial Intelligence; Intensive Care Unit
MeSH Terms: interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with carbapenem resistant Klebsiella spp. infection
  Interventions: Other: Artificial intelligence
- Patients with carbapenem sensitive Klebsiella spp. infection
  Interventions: Other: Artificial intelligence

INTERVENTIONS:
Other: Artificial intelligence — Prediction of carbapenem resistance via deep machine learning model

SUMMARY:
The aim of this study to predict carbapenem resistant Klebsiella spp. earlier in our patients monitored in our Intensive Care Unit in the future, using artificial intelligence.

Patients with bloodstream infection and pneumonia caused by Klebsiella spp. will be comparatively examined in two groups, as sensitive and resistant. Resistance will be attempted to be predicted with deep machine learning.

DETAILED DESCRIPTION:
Antimicrobial resistance is a globally increasing threat and has serious consequences on both public health and the economy. In an infection that may develop with a resistant microorganism, therapeutic options are limited, hence early and effective treatment that can be initiated by predicting resistance will make a difference in patient prognosis.

Today, artificial intelligence and machine learning are changing our medical practice. When the literature is reviewed, there are studies suggesting that machine learning can predict antimicrobial resistance.Risk factors for carbapenem-resistant Klebsiella spp. have been previously identified. These previously identified risk factors will be evaluated retrospectively in our own patients and an algorithm related to the prediction of resistance will be developed with the help of machine learning.

Our goal is to predict bacterial resistance earlier in our patients monitored in our Intensive Care Unit in the future, using artificial intelligence, and to facilitate our patients' access to early and effective treatment options.

Secondarily, it is also aimed to provide economic benefits by preventing unnecessary antibiotic use.

Access to patients' data will be obtained retrospectively through the hospital automation system.

Publications in the literature will be examined, and the risk factors causing the development of infection with carbapenem-resistant Klebsiella spp. will be evaluated.

Patients with carbapenem resistance and sensitivity will be compared in two separate subgroups.

The obtained features will be classified using various decision trees and neural algorithms separately. The data obtained will be statistically compared in the distinction of resistance and sensitivity. Statistical evaluation was done with IBM SPSS 29.0 (IBM Corp., Armonk, NY, USA). Demographic data, descriptive statistics, Categorical variables will be expressed in terms of frequency (percentage).

Categorical variables will be expressed with the chi-square test. The performance of Machine Learning algorithms will be evaluated by ROC analysis, AUC, classification accuracy, sensitivity, and specificity values will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Patients monitored in our third-level intensive care unit between June 2017 and June 2023 will be evaluated retrospectively. Patients with pneumonia and bloodstream infection developed with Klebsiella spp. will be included in the study.

Exclusion Criteria:

* Patients under the age of 18 have not been included in the study.
* Infections outside of the respiratory tract and bloodstream have not been included in the study.
* Patients with respiratory tract colonization and without active inflammation have also not been included.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients monitored in our third-level intensive care unit between June 2017 and June 2023 will be evaluated retrospectively. Patients with pneumonia and bloodstream infection developed with Klebsiella spp. will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Risk of Carbapenem Resistant Klebsiella Infection | 3 months
  The sensitivity and specificity of a diagnostic method based on machine learning will be measured with the AUC-ROC curve (Area Under the Receiver Operating Characteristic curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alparslan V, Guler O, Inner B, Duzgun A, Baykara N, Kus A. A novel approach to antimicrobial resistance: Machine learning predictions for carbapenem-resistant Klebsiella in intensive care units. Int J Med Inform. 2025 Mar;195:105751. doi: 10.1016/j.ijmedinf.2024.105751. Epub 2024 Dec 7. PMID 39674007
- See also: Using Machine Learning to Predict Antimicrobial Resistance of Acinetobacter Baumannii, Klebsiella Pneumoniae and Pseudomonas Aeruginosa Strains — https://pubmed.ncbi.nlm.nih.gov/34042702/